CLINICAL TRIAL: NCT00925535
Title: Open-Label, Randomized, 3-Way Crossover Study To Estimate The Interaction Between Multiple Dose Rifabutin And Lersivirine (UK-453,061) In Healthy Subjects
Brief Title: Drug Interaction Study Between Rifabutin And Lersivirine (UK-453,061)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A5271043
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics HIV Tuberculosis Lersivirine UK-453; 061 Rifabutin; HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — UK 453,061; Rifabutin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Active Comparator): Lersivirine
  Interventions: Drug: Lersivirine
- Treatment B (Active Comparator): Rifabutin
  Interventions: Drug: Rifabutin
- Treatment C (Experimental): Lersivirine and Rifabutin
  Interventions: Drug: Lersivirine; Drug: Rifabutin

INTERVENTIONS:
Drug: Lersivirine — 1000 mg once daily for 10 days
  Arms: Treatment A
Drug: Rifabutin — 300 mg once daily for 10 days
  Arms: Treatment B
Drug: Lersivirine — 1000 mg once daily for 10 days
  Arms: Treatment C
Drug: Rifabutin — 300 mg once daily for 10 days
  Arms: Treatment C

SUMMARY:
Approximately 1/3 of persons living with HIV infection are co-infected with tuberculosis (TB). Rifabutin, used in the treatment of TB, is an inducer of drug metabolism thus may decrease concentrations of lersivirine if co-administered. Lersivirine is a modest inducer of drug metabolism, thus lersivirine may decrease concentrations of rifabutin as well.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* History of regular alcohol consumption exceeding 7 drinks/week for women and 14 drinks/week for men (1 drink = 150 mL of wine or 360 mL of beer or 45 mL of hard liquor).
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.
* Hypersensitivity/allergic reactions to any component of the study drugs.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Lersivirine plasma pharmacokinetic parameters: AUC24, Cmax, Tmax, and C24h | 20 days
Rifabutin and 25-O-desacetyl-rifabutin plasma pharmacokinetic parameters: AUC24, Cmax, Tmax, and C24h | 20 days

SECONDARY OUTCOMES:
Safety and toleration assessed by spontaneous reporting of adverse events, vital signs, 12 lead ECG and laboratory safety assessments | 58 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5271043&StudyName=Drug%20Interaction%20Study%20Between%20Rifabutin%20And%20Lersivirine%20%28UK-453%2C061%29